CLINICAL TRIAL: NCT03366402
Title: Sub Populations of Immune Cells in Influenza A and B Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Nechama Sharon (Other)
Responsible Party: Sponsor-Investigator, Dr. Nechama Sharon, Head of Pediatric Hemato-Oncology Unit, Depute Director Department of Pediatrics, Laniado Hospital
Organization: Laniado Hospital (Other)
Other Study IDs: 0015-16-LND
Record Dates: First submitted 2017-11-16; First posted 2017-12-08 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Influenza A and B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Influenza A
  Interventions: Diagnostic Test: RT-PCR H1N1
- Influenza B
  Interventions: Diagnostic Test: RT-PCR H1N1

INTERVENTIONS:
Diagnostic Test: RT-PCR H1N1 — At the first stage an upper respiratory swab was taken to determine the presence of Infuenza A H1N1 (the virus identification was done by RT - PCR). Then the different subtypes of lymphocytes were quantified at different stages of the disease. The identification and quantification of the different cell types were performed by FACS method, the cell receptors that were marked were CD31, CD19, CD4, CD3, CD45, CD8, CD56.

SUMMARY:
This study designed to examine changes of immune system cells sub-populations during influenza disease. Several parameters will be examined, such as: amount of sub populations, clinical parameters (body temperature and number of hospitalization days).

The participants are children that are hospitalized in the Laniado hospital pediatric department.

DETAILED DESCRIPTION:
Background:

In late March and early April 2009 an outbreak of a novel influenza virus designated A/H1N1 influenza (popularly known as swine flu) was reported in Mexico, with subsequent cases observed in many countries, leading to the declaration by the World Health Organization of a worldwide pandemic.

The first case of influenza A/H1N1 in Israel was diagnosed at the end of April 2009 at Laniado Hospital in a young man returning from Mexico.

Influenza A/H1N1 (Swine flu) carries a relatively high morbidity, particularly in young patients. Early identification would enable prompt initiation of therapy, thereby improving outcomes.

In 2009, during the H1N1 pandemic in Israel, a research was conducted in our department of pediatrics. The researchers Sharon et al. (1) have compared a group of 53 children infected with Influenza A H1N1, with a group of 53 children that presented with flu symptoms but were found negative for the virus. This comparison demonstrated a significant reduction in lymphocyte count during the acute phase of the disease (days 1-3) with resolution on day 7 (6-9) as well as reduction in the neutrophil count on day 5 from the onset of high fever with subsequent resolution 2-4 days later (days 7-10). This phenomenon was not observed in the patients that were not infected with the H1N1 virus. Similar results were reported by Cao and co-authors (2) that observed it in both pediatric and adult patients. Lewis at al suggested that the lymphopenia is mainly due to reduction in T cells and to a lesser extent in B cells (3). The lymphopenia typical of influenza A H3N3 during acute illness was shown to be due to a reduction in both T and B cells without alteration in the CD4:CD8 ratio. This is in contrast to the findings of Cao et al. (2) who noted an abnormal CD4:CD8 ratio in half of those who were positive for A H1N1. One of the possible explanations as proposed by Nichols and Collaborators (4) is that early lymphopenia and the later neutropenia in the influenza infected patients may represent migration of these cells from the circulation to the infected respiratory tract as a consequence of infection. Goals of our research To quantify the B, T and NK populations of lymphocytes during different stages of the disease caused by Infuenza A H1N1.

Study methods The subjects of the study were children that were hospitalized at our department with signs and symptoms of flu. The parents or legal guardians of the participants have signed a written consent. At the first stage an upper respiratory swab was taken to determine the presence of Infuenza A H1N1 (the virus identification was done by RT - PCR). Then the different subtypes of lymphocytes were quantified at different stages of the disease. The identification and quantification of the different cell types were performed by FACS method, the cell receptors that were marked were CD31, CD19, CD4, CD3, CD45, CD8, CD56.

Laboratory technique:

Cellular markers were assessed by flow cytometry. Cell staining was performed on single cell suspensions using pre-cooled PBS in 5 ml FACS tubes. Washing steps were performed by centrifugation for 5min, 300 g, 5°C, brake 5 after which supernatants were completely pipetted off and cell pellets (typically containing 0.2-1.0×106 cells) were re-suspended in 100 μl PBS (without Ca++and Mg++) supplemented with 0.5% bovine serum albumin, stained with specific fluorochrome-conjugated anti-human antibodies or isotype-matched non-specific controls and incubated in the refrigerator 2-8°C for 30 min. After incubation, cells were washed by centrifugation and re-suspended in 0.25-0.5 ml cold PBS.

Cells tested were stained with mouse monoclonal antibodies for CD45-FITC, CD45-PE a pan leukocyte marker, T Cell marker CD3-PE CD8-FITC, T helper cells CD4-FITC, CD8-PE, Natural killer (NK) cell marker CD56-PE, monocyte marker CD31-FITC and B cell marker CD19-PE.

Emission compensation was done by positive control tubes containing cells that were stained with CD45-FITC or CD45-PE; Dead cells were excluded by staining with 7-aminoactinomycin D, only un-stained viable cells were analyzed. At least 10,000 cellular events per sample were analyzed using the CellQuest Pro or FlowJo software. Percentages of isotype control antibody staining, not exceeding 1% stained cells, were used to set the 'positive'staining gates, and were deduced from the specific antibody results. The results are expressed as the percentage of stained cells.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-16
* Have signed a written consent by parents or legal guardians
* Signs and symptoms of flu

Exclusion Criteria:

* Immune system disease

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalized at the pediatric department with signs and symptoms of flu.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Quantifing the B, T and NK populations of lymphocytes during different stages of the disease caused by Infuenza A H1N1. | 2 years
  The identification and quantification of the different cell types are performed by FACS method, the cell receptors that were marked were CD31, CD19, CD4, CD3, CD45, CD8, CD56.
  The primary outcome measure was defined as the absolute number of lymphocytes of each sub population. Thus, farther allowing us to follow both absolute numbers and relative percentage of the whole.

CONTACTS AND LOCATIONS:
Locations (1):
- Sharon Nechama, Laniado Hospital, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No